CLINICAL TRIAL: NCT02898584
Title: Utilizing Consumer Health Informatics to Support Management of Hypertension by Clinical Pharmacists in Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Lorraine Buis, Assistant Professor of Family Medicine, Medical School and Assistant Professor of Information, School of Information, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MICHR T3-RIP; HUM00105772 (Other: University of Michigan)
Record Dates: First submitted 2016-09-08; First posted 2016-09-13 (Estimated); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BP Track (Other): The study participants will be asked to monitor their blood pressure twice daily at home for twelve weeks, and sync the data to the mobile intervention so that a clinical pharmacist can review and incorporate the data into ongoing hypertension management.
  Interventions: Other: BP Track

INTERVENTIONS:
Other: BP Track

SUMMARY:
The purpose of this research study is to test the feasibility, acceptability, and preliminary effectiveness of the use of a mobile pharmacist-led intervention that incorporates home BP monitoring and medication reminders with patients recruited from a primary care setting, as well as identify challenges and potential solutions to broader implementation of a mobile pharmacist-led home-based BP monitoring intervention in primary care clinics through key stakeholder interviews.

ELIGIBILITY:
Inclusion Criteria:

* Have a smart phone compatible with mobile intervention
* Have been previously diagnosed with hypertension
* Have uncontrolled hypertension (systolic blood pressure > 140 and/or diastolic blood pressure > 90 on repeat measurement)
* Be under the care of a primary care physician at the recruitment clinic
* Be taking at least one antihypertensive medication
* Be English speaking

Exclusion Criteria:

* Patients under the care of a clinical pharmacist for hypertension management, or under the care of a cardiologist
* Pregnant patients and anyone with the following unrelated, but serious medical conditions will also be excluded, as they may make blood pressure control difficult or necessitate frequent hospitalization: previous diagnosis of resistant hypertension; steroid dependent asthma or emphysema; cirrhosis or hepatic failure; stage C or D chronic heart failure; stage IV or V chronic kidney disease; and cancer (terminal or undergoing active chemotherapeutic or radiation therapy)
* Patients with other serious medical conditions (e.g., stroke, dementia) that may affect their ability to self-monitor blood pressure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-10; Primary Completion 2020-06 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | from baseline to 12 weeks

SECONDARY OUTCOMES:
Change in medication adherence as measured by the Adherence to Refills and Medications Scale (ARMS) | from baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lorraine R Buis, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Buis LR, Roberson DN, Kadri R, Rockey NG, Plegue MA, Danak SU, Guetterman TC, Johnson MG, Choe HM, Richardson CR. Understanding the Feasibility, Acceptability, and Efficacy of a Clinical Pharmacist-led Mobile Approach (BPTrack) to Hypertension Management: Mixed Methods Pilot Study. J Med Internet Res. 2020 Aug 11;22(8):e19882. doi: 10.2196/19882. PMID 32780026
- [Derived] Buis LR, Roberson DN, Kadri R, Rockey NG, Plegue MA, Choe HM, Richardson CR. Utilizing Consumer Health Informatics to Support Management of Hypertension by Clinical Pharmacists in Primary Care: Study Protocol. JMIR Res Protoc. 2017 Oct 10;6(10):e193. doi: 10.2196/resprot.8059. PMID 29017994